CLINICAL TRIAL: NCT05625724
Title: Aspirin for the Prevention of Preeclampsia and Pregnancy Outcomes in Nulliparous Women After Assisted Reproductive Technology. APPART
Brief Title: Aspirin for the Prevention of Preeclampsia and Pregnancy Outcomes After Assisted Reproductive Technology
Acronym: APPART
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC31/21/0337
Record Dates: First submitted 2022-11-14; First posted 2022-11-23 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: ART; Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): Low-dose Aspirin: 150mg, daily, oral route, at bedtime, initiated between 9 and 14 weeks of gestation, until 35 (+6) weeks of gestation, or in the event of earlier delivery, until the onset of labor.
  Interventions: Drug: Aspirin
- Control (Placebo Comparator): Matching placebo administrated daily, oral route, at bedtime, initiated between 9 and 14 weeks of gestation, until 35 (+6) weeks of gestation, or in the event of earlier delivery, until the onset of labor.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Experimental drug administrated orally
  Arms: Aspirin
Drug: Placebo — Treatment for the control group
  Arms: Control

SUMMARY:
This study seeks to validate the hypothesis that nulliparous pregnant women after Assisted Reproductive Technology (ART) are at high risk of preeclampsia and perinatal complications and represent a subgroup for which aspirin prophylaxis during pregnancy may be effective in the prevention of preterm preeclampsia and other perinatal adverse outcomes.

DETAILED DESCRIPTION:
Preeclampsia (PE) affects 2% of pregnancies in France and is an important cause of maternal and perinatal mortality and morbidity. Aspirin is currently the only prophylactic therapy for PE in high-risk women when initiated before 16 weeks of gestation and at a daily dose of 100-160 mg, with a reduction in the incidence of preterm preeclampsia of 60-70% in recent meta-analysis. Latest data also demonstrate a potential beneficial effect of aspirin on spontaneous preterm birth. A major challenge in modern obstetrics is early identification of pregnant women at high-risk of PE who could benefit from aspirin treatment. In France, the College National des Gynécologues et Obstétriciens Français and the Société Française d'HyperTension Artérielle have restrictive recommendation of aspirin to be prescribed only to women with a history of PE or vascular intra-uterine growth restriction, thus leaving out all nulliparous women (including those with multiple risk factors). Other countries (USA, United Kingdom (UK), Canada) have much broader recommendations with aspirin prescription for patients with one high or 2 moderate risk factors, but exposing nearly 30% of pregnant women to aspirin (leading to unnecessary exposure to treatment). The Fetal Medicine Foundation provides a screening test combining clinical parameters, uterine artery Doppler, and biomarkers; but this strategy has high false-positive rate and the reproducibility needs to be confirmed in clinical practice.

It seems necessary to be able to better target women at risk, especially in nulliparous women. Nulliparity and assisted reproductive technology (ART) are independent risk factors for PE. Currently the proportion of pregnancy after ART in France is roughly 6.9% and is rising. Nulliparous ART pregnant women have a higher risk of PE and preterm birth. Indeed, they commonly cumulate risk factors including age>35years in association with nulliparity and ART. The rate of PE in this population can rise up to 10%.

Our hypothesis is that nulliparous pregnant women after ART are at high risk of preeclampsia and perinatal complications and represent a subgroup for which aspirin prophylaxis during pregnancy may be effective in the prevention of preterm preeclampsia and other perinatal adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women aged 18 years or more
* Pregnancy following ART, including in vitro fertilization (IVF), intracytoplasmic sperm injection (ICSI), oocyte donation or intrauterine insemination with sperm donor
* Singleton pregnancy
* Evolutive pregnancy between 9 and 14 weeks of gestation
* Women affiliated to a French Social Security Insurance or equivalent social protection
* Written informed consent

Exclusion Criteria:

* Major fetal abnormality
* Regular treatment with aspirin (including antiphospholipid syndrome)
* Aspirin contraindications (allergy, von Willebrand disease, peptic ulceration, hemophilia)
* Women protected by law.
* Women included in another interventional study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo in the prevention of preterm (<37 weeks of gestation) preeclampsia | Up to 9 months
  Occurrence of preterm (<37 weeks of gestation) preeclampsia (binary variable yes/no)

SECONDARY OUTCOMES:
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on spontaneous and total preterm birth <34 weeks of gestation | Up to 8 months
  Occurrence of spontaneous and total preterm birth (defined by delivery at <34 weeks of gestation)
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on spontaneous and total preterm birth <37 weeks of gestation | Up to 9 months
  Occurrence of spontaneous and total preterm birth (defined by delivery at <37weeks of gestation)
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on occurrence of preeclampsia <34 weeks of gestation, term preeclampsia (≥ 37 weeks of gestation) | Up to 8 months
  Occurrence of term (≥37 weeks) preeclampsia
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on occurrence of cesarean delivery | Up to 9 months
  Occurrence of cesarean delivery
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on occurrence of postpartum hemorrhage (>500ml) | Up to 9 months
  Occurrence of postpartum hemorrhage (>500ml)
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on occurrence of placental abruption | Up to 9 months
  Occurrence of placental abruption
Compare the effect of aspirin 150mg daily initiated between 9 and 14 weeks of gestation versus placebo on neonatal adverse outcome. | Up to 9 months
  Occurrence of neonatal adverse outcomes: still birth, neonatal death, neonatal complications

CONTACTS AND LOCATIONS:
Overall Officials: Christophe VAYSSIERE, MD, Principal Investigator — University Hospital, Toulouse
Locations (21):
- France (21):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon-Bourgogne, Dijon
  - CHU Lille, Lille
  - HCL - Groupement Hospitalier Est, Hôpital Femme Mère Enfant, Lyon
  - AP-HM Hôpital de la Conception, Marseille
  - AP-HM Hôpital Nord, Marseille
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nîmes, Nîmes
  - Groupe hospitalier St Joseph, Paris
  - Hôpital Armand - Trousseau, Paris
  - Hôpital Cochin, Paris
  - CHI Poissy Saint Germain en Laye, Poissy
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Saint Etienne, Hôpital Nord, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No